CLINICAL TRIAL: NCT02163993
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled Study of Galcanezumab in Patients With Episodic Migraine
Brief Title: A Study of Galcanezumab (LY2951742) in Participants With Migraine Headache
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15414; I5Q-MC-CGAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2017-06

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 5mg Galcanezumab (Experimental): 5mg of galcanezumab given as subcutaneous (SQ) injections once every 28 days during a 12 week treatment period.
  Interventions: Drug: Galcanezumab
- 50mg Galcanezumab (Experimental): 50mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
  Interventions: Drug: Galcanezumab
- 120mg Galcanezumab (Experimental): 120mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
  Interventions: Drug: Galcanezumab
- 300mg Galcanezumab (Experimental): 300mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo given as SQ injections once every 28 days during a 12 week treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SQ
  Other Names: LY2951742
  Arms: 120mg Galcanezumab; 300mg Galcanezumab; 50mg Galcanezumab; 5mg Galcanezumab
Drug: Placebo — Administered SQ
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate whether the study drug known as galcanezumab is safe and effective in the prevention of migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a history of migraine of at least 1 year prior to enrollment.
* Migraine onset prior to age 50.

Exclusion Criteria:

* Current enrollment in, or discontinuation within the last 30 days from, a clinical trial involving any investigational drug or device.
* Current use or any prior exposure to any CGRP antibody, any antibody to the CGRP receptor, or antibody to nerve growth factor (NGF).
* History of migraine subtypes including hemiplegic migraine, ophthalmoplegic migraine, and basilar-type migraine.
* Have a history or presence of other medical illness that indicates a medical problem that would preclude study participation.
* Failure to respond to more than two adequately dosed effective migraine prevention treatments.
* Evidence of significant active psychiatric disease, in the opinion of the investigator.
* Women who are pregnant or nursing.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2015-08-19 (Actual); Study Completion 2018-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (40):
  - Clinical Research Advantage, Gilbert, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Pharmacology Research Institute, Long Beach, Encino, California
  - Collaborative Neuroscience Network - CNS, Long Beach, California
  - Pharmacology Research Institute, Long Beach, Los Alamitos, California
  - Pharmacology Research Institute, Long Beach, Newport Beach, California
  - Desert Valley Research, Rancho Mirage, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - New England Institute for Clinical Research, Stamford, Connecticut
  - Avail Clinical Research LLC, DeLand, Florida
  - Florida Clinical Research Center LLC, Maitland, Florida
  - Renstar Medical Research, Ocala, Florida
  - Psychiatric Inst of Florida-Clinical Neuroscience Solutions, Orlando, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Otri-Med Corporation, Edgewood, Kentucky
  - PharmaSite Research Inc, Baltimore, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Westside Family Medical Center, Kalamazoo, Michigan
  - ClinVest, Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Island Neuro Associates,PC, Plainview, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - PharmQuest, Greensboro, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Summit Research Network Inc, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - CNS Health Care, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
  - DermResearch, Austin, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
  - North Seattle Womens Group, Seattle, Washington
  - Dean Foundation for Health Research and Education, Middleton, Wisconsin

REFERENCES:
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Bangs ME, Kudrow D, Wang S, Oakes TM, Terwindt GM, Magis D, Yunes-Medina L, Stauffer VL. Safety and tolerability of monthly galcanezumab injections in patients with migraine: integrated results from migraine clinical studies. BMC Neurol. 2020 Jan 17;20(1):25. doi: 10.1186/s12883-020-1609-7. PMID 31952501
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569
- [Derived] Skljarevski V, Oakes TM, Zhang Q, Ferguson MB, Martinez J, Camporeale A, Johnson KW, Shan Q, Carter J, Schacht A, Goadsby PJ, Dodick DW. Effect of Different Doses of Galcanezumab vs Placebo for Episodic Migraine Prevention: A Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):187-193. doi: 10.1001/jamaneurol.2017.3859. PMID 29255900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment period (0 to 12 weeks), Post-treatment period (12 to 24 weeks)
Groups:
- Placebo: Placebo given as subcutaneous (SQ) injections once every 28 days during a 12 week treatment period.
- 5mg Galcanezumab: 5mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
Period: Treatment Period
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Started | 138 | 68 | 68 | 71 | 69
Received at Least 1 Dose of Study Drug | 137 | 68 | 68 | 70 | 67
Completed | 126 | 59 | 66 | 62 | 62
Not Completed | 12 | 9 | 2 | 9 | 7
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1 | 3 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 6 | 4 | 1 | 4 | 1
Not completed — Not treated | 1 | 0 | 0 | 1 | 2
Period: Post-treatment Period
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Started | 125 (One participant discontinued after Treatment Period. Did not enter into Post-treatment Period.) | 61 (Participants who discontinued or completed the Treatment Period entered the Post-treatment period.) | 66 | 63 (Participants who discontinued or completed the Treatment Period entered the Post-treatment period.) | 65 (Participants who discontinued or completed the Treatment Period entered the Post-treatment period.)
Completed | 121 | 55 | 62 | 61 | 62
Not Completed | 4 | 6 | 4 | 2 | 3
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 3 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab | Total
Number analyzed (Participants) | 137 | 68 | 68 | 70 | 67 | 410
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.54 (12.10) | 41.40 (11.15) | 39.63 (12.42) | 40.57 (10.92) | 40.79 (13.20) | 40.24 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 55 | 61 | 59 | 56 | 340
  Male | 28 | 13 | 7 | 11 | 11 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 14 | 11 | 8 | 14 | 67
  Not Hispanic or Latino | 117 | 54 | 57 | 62 | 53 | 343
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 0 | 2
  Asian | 6 | 1 | 0 | 3 | 1 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 16 | 9 | 23 | 13 | 75
  White | 106 | 49 | 57 | 43 | 52 | 307
  More than one race | 9 | 2 | 2 | 1 | 1 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 137 | 68 | 68 | 70 | 67 | 410
Number of migraine headache days [Mean (Standard Deviation); unit: Days] — Migraine Headache Day: A calendar day on which a migraine headache occurred.
  Days | 6.64 (2.73) | 6.68 (2.73) | 6.41 (2.66) | 6.95 (2.56) | 6.73 (2.48) | 6.68 (2.64)
Number of probable and migraine headache days [Mean (Standard Deviation); unit: Days] — Probable Migraine Headache Day: A calendar day on which a probable migraine headache occurred.
  Days | 8.04 (3.08) | 8.55 (3.23) | 8.33 (3.21) | 8.69 (3.46) | 8.01 (2.79) | 8.28 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Number of Migraine Headache Days in the Last 28-Day Period of the 12-Week Treatment Phase
Description: The criteria for a migraine headache was adapted from the standard International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta. The definition of a migraine headache was a headache with or without aura, of ≥30 minutes (min) duration, and with both ("A" and "B") required features from the IHS ICHD-3 beta definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia.
Time Frame: Baseline, 12 Weeks
Population: All participants with a valid 28-day baseline assessment of migraine headache days who received at least 1 dose of study treatment and had evaluable postbaseline headache data.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Days | -3.66 (0.28) | -4.23 (0.37) | -3.92 (0.36) | -4.80 (0.37) | -4.28 (0.39)
Statistical Analysis 1: Comparison: Placebo vs 5mg Galcanezumab; Test type: Superiority; Bayesian Dose Response Model; Posterior Mean Difference = -0.57, 95% CI 2-sided [-1.40 to 0.24], Standard Deviation 0.42
Statistical Analysis 2: Comparison: Placebo vs 50mg Galcanezumab; Test type: Superiority; Bayesian Dose Response Model; Posterior Mean Difference = -0.25, 95% CI 2-sided [-1.06 to 0.56], Standard Deviation 0.41
Statistical Analysis 3: Comparison: Placebo vs 120mg Galcanezumab; Test type: Superiority; Bayesian Dose Response Model; Posterior Mean Difference = -1.14, 95% CI 2-sided [-2.02 to -0.29], Standard Deviation 0.44
Statistical Analysis 4: Comparison: Placebo vs 300mg Galcanezumab; Test type: Superiority; Bayesian Dose Response Model; Posterior Mean Difference = -0.62, 95% CI 2-sided [-1.50 to 0.27], Standard Deviation 0.45

2. Secondary Outcome: Mean Change From Baseline in Number of Migraine Attacks in the Last 28-Day Period of the 12-Week Treatment Phase
Description: A migraine attack was defined as beginning on any day a migraine headache day was recorded and ending when a migraine headache-free day occurred. The criteria was adapted from the standard IHS ICHD-3 beta definition. The definition of a migraine headache was a headache with or without aura, of ≥30 minutes (min) duration, and with both ("A" and "B") required features from the IHS ICHD-3 beta definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia. Least Squares (LS) mean was calculated using mixed model repeated measures (MMRM) methodology with treatment, pooled investigative site, period, and treatment-by-period interaction, baseline and baseline-by-period interaction.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Migraine attacks
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Migraine attacks | -2.65 (0.17) | -2.98 (0.23) | -2.87 (0.22) | -3.46 (0.23) | -3.01 (0.23)

3. Secondary Outcome: Percentage of Participants With ≥50% Reduction in Number of Migraine Headache Days in the Last 28-Day Period of the 12-Week Treatment Phase
Description: The criteria for a migraine headache was adapted from the standard International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta definition. The definition of a migraine headache was a headache with or without aura, of ≥30 minutes (min) duration, and with both ("A" and "B") required features from the IHS ICHD-3 beta definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia.
Time Frame: Week 12
Population: All participants with a valid 28-day baseline assessment of migraine headache days who received at least 1 dose of study treatment and had evaluable postbaseline headache data during the time period of analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Percentage of participants | 60.9 | 75.4 | 65.5 | 76.5 | 70.1

4. Secondary Outcome: Mean Change From Baseline in the Number of Days of Medication Use for the Treatment of Migraine Headache in the Last 28-Day Period of the 12-Week Treatment Phase
Description: A migraine attack was defined as beginning on any day a migraine headache day was recorded and ending when a migraine headache-free day occurred. The criteria was adapted from the standard IHS ICHD-3 beta definition. The definition of a migraine headache was a headache with or without aura, of ≥30 minutes (min) duration, and with both ("A" and "B") required features from the IHS ICHD-3 beta definition. Required feature "A" includes at least 2 of the following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of the following during the headache: nausea and/or vomiting, or photophobia and phonophobia. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with treatment, pooled investigative site, period, and treatment-by-period interaction, baseline and baseline-by-period interaction.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Days | -2.51 (0.23) | -3.27 (0.32) | -2.58 (0.31) | -3.59 (0.31) | -3.15 (0.32)

5. Secondary Outcome: Mean Change From Baseline in Number of Headache Hours in the Last 28-Day Period of the 12-Week Treatment Phase
Description: Number of headache hours calculated as the total number of headache hours in a 28-day period on which a headache occurred. Least Squares (LS) means was determined by mixed model repeated measures (MMRM) methodology with treatment, pooled investigative site, period, and treatment-by-period interaction, baseline and baseline-by-period interaction.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Hours | -16.56 (1.73) | -20.15 (2.45) | -19.38 (2.35) | -22.29 (2.39) | -24.45 (2.42)

6. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Migraine Specific Quality of Life (MSQL) Questionnaire Total Scores
Description: MSQL consists of 14 questions across 3 dimensions (role function-restrictive, role function-preventive, and emotional function). All question values range from 1 to 6. Participants rated each item from 1 (none of the time) to 6 (all of the time). Since each item was presented as a negative statement, participant responses were recorded before item scores were calculated. Then, dimension scores were calculated as the sum of the recorded items for that specific dimension. Each dimension score was transformed into a score that ranged from 0 to 100. The transformation formula for the restrictive function = [(dimension score-7)*100]/35, for the preventive function = [(dimension score-4)*100]/20, and for the emotional function = [(dimension score-3)*100]/15. A lower score indicated a poorer quality of life associated with that domain. LS means was determined by Analysis of covariance (ANCOVA) with treatment, pooled investigative site and baseline.
Time Frame: Baseline, 12 Weeks
Population: All randomized participants who received at least 1 dose of study drug and have non-missing values at baseline and post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 133 | 63 | 67 | 63 | 64
units on a scale | 21.08 (1.82) | 27.53 (2.53) | 25.35 (2.46) | 30.23 (2.58) | 27.49 (2.51)

7. Secondary Outcome: Change From Baseline to 12 Week Endpoint in the Headache Impact Test-6™ (HIT-6™) Scores
Description: The HIT-6 consists of 6 questions to measure the impact of headaches on the participants ability to function on the job, at school, at home and in social situations. A score to each question will be assigned as follows: never - 6, rarely - 8, sometimes - 10, very often - 11, and always - 13. The composite score is calculated as the sum of the scores for all 6 questions, the total score ranges between 36 and 78 with higher total scores reflecting more severe impact of headaches. LS means was determined by ANCOVA with treatment, pooled investigative site and baseline.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 133 | 63 | 67 | 63 | 64
units on a scale | -7.26 (0.79) | -9.26 (1.09) | -8.46 (1.06) | -9.95 (1.12) | -8.27 (1.09)

8. Secondary Outcome: Serum Concentration of Galcanezumab
Description: Blood serum concentrations of galcanezumab.
Time Frame: 12 Weeks
Population: All randomized participants who received at least 1 dose of study drug with non-missing baseline and postbaseline measures for serum concentration of galcanezumab.
Measure: Mean (Standard Deviation); unit: nanomoles per litre (nmol/L)
Arm/Group | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 59 | 66 | 62 | 63
nanomoles per litre (nmol/L) | 840 (602) | 4650 (2430) | 13200 (7060) | 32100 (19100)

9. Secondary Outcome: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: CGRP has been shown to be involved in the pathophysiology of migraine through dilation of cerebral and dural blood vessels, release of inflammatory mediators, and transmission of nociceptive (pain) information from intracranial blood vessels to the nervous system (Villalón and Olesen 2009). In migraineurs, serum concentrations of CGRP are significantly elevated during migraine attacks (Goadsby et al. 1990; Goadsby and Edvinsson 1993).
Time Frame: 12 Weeks
Population: All randomized participants who received at least 1 dose of study drug with non-missing baseline and postbaseline measures for CGRP plasma concentration.
Measure: Mean (Standard Deviation); unit: nanomoles per litre (nmol/L)
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 14 | 55 | 63 | 61 | 63
nanomoles per litre (nmol/L) | 0.1810 (0.1030) | 0.4750 (0.3940) | 1.5700 (0.7010) | 2.8000 (1.2200) | 3.8300 (1.3100)

10. Secondary Outcome: Percentage of Participants Developing Anti-drug Antibodies to Galcanezumab
Description: The percent of participants with treatment emergent Anti-drug Antibodies (ADA) were assessed at week 1 to 12. A participant was considered to have treatment-emergent Galcanezumab ADA if the participant had at least 1 titer that was treatment-emergent relative to baseline, defined as any of the following: A negative baseline ADA result and a subsequent positive post-baseline ADA result with a titer >=20; or a positive ADA results and a subsequent positive post-baseline ADA results with a 4-fold or greater increase in titer from the baseline measurement.
Time Frame: Baseline through 12 Weeks
Population: All randomized participants who received at least 1 dose of study drug with non-missing baseline and postbaseline ADA measures.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 136 | 65 | 66 | 68 | 65
Percentage of participants | 2.2 | 7.7 | 4.6 | 2.9 | 3.1

11. Secondary Outcome: Percentage of Participants With Suicidal Ideation and Behaviors Assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) Scores
Description: The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal behavior: a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide.
Time Frame: Baseline through Week 12
Population: All randomized participants who received at least 1 dose of study drug and with non-missing baseline and postbaseline C-SSRS assessment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 136 | 66 | 67 | 68 | 66
Percentage of Participants
  Suicidal Ideation | 0 | 0 | 0 | 0 | 1.52
  Suicidal Behavior | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Mean Change From Baseline in the Number of Headache Days in the Last 28-Day Period of the 12-Week Treatment Phase
Description: Number of calendar days on which a headache lasts ≥4 hours which includes migraines, probable migraines (PM) and nonmigraines. Criteria for migraine headache (MH) was adapted from standard IHS ICHD-3 beta definition. It is defined as headache with or without aura, of ≥30 min duration, and with both ("A" and "B") required features from IHS ICHD-3 beta definition. Required feature "A" includes ≥2 of following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of following during headache: nausea and/or vomiting, or photophobia and phonophobia. PM is headache with or without aura, but missing 1 feature needed to fulfill all criteria for MH. LS means were calculated using MMRM with treatment, pooled investigative site, period, and treatment-by-period interaction, baseline and baseline-by-period interaction.
Time Frame: Baseline, 12 Weeks
Population: All randomized participants with a valid 28-day baseline assessment of migraine headache days who received at least 1 dose of study treatment and had evaluable postbaseline headache data.
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Days | -2.47 (0.22) | -2.81 (0.32) | -2.57 (0.30) | -3.11 (0.31) | -3.37 (0.31)

13. Secondary Outcome: Mean Change From Baseline in the Number of Moderate-Severe Headache Days in the Last 28-Day Period of the 12-Week Treatment Phase
Description: Number of calendar days on which headache lasts ≥4 hrs it includes migraines, PM & non-migraines. MH is headache with or without aura, of ≥30 min duration, and with both ("A" and "B") required features from IHS ICHD-3 beta definition. Required feature "A" includes ≥2 of following headache characteristics: unilateral location, pulsatile quality, moderate or severe pain intensity, or aggravation by or causing avoidance of routine physical activity. Required feature "B" includes at least 1 of following during headache: nausea &/or vomiting, or photophobia & phonophobia. PM is headache with or without aura, but missing 1 feature needed to fulfill all criteria for MH. Severity was measured via interactive voice response system questionnaire "What was the worst headache pain? For mild press 1. For moderate 2. For severe press 3". LSmean was calculated using MMRM with treatment, pooled investigative site, period, treatment-by-period interaction, baseline and baseline-by-period interaction.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Placebo | 5mg Galcanezumab | 50mg Galcanezumab | 120mg Galcanezumab | 300mg Galcanezumab
Number analyzed (Participants) | 134 | 65 | 68 | 69 | 66
Days | -2.33 (0.20) | -2.49 (0.28) | -2.33 (0.27) | -2.88 (0.28) | -3.13 (0.28)

ADVERSE EVENTS:
Time Frame: Up To 24 Weeks
Groups:
- Placebo - Treatment Phase; Placebo - Post-Treatment Phase: Placebo given as SQ injections once every 28 days during a 12 week treatment period.
- 5mg Galcanezumab-Treatment Phase; 5mg Galcanezumab-Post-Treatment Phase: 5mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
- 50mg Galcanezumab-Treatment Phase; 50mg Galcanezumab-Post-Treatment Phase: 50mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
- 120mg Galcanezumab-Treatment Phase; 120mg Galcanezumab-Post-Treatment Phase: 120mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
- 300mg Galcanezumab-Treatment Phase; 300mg Galcanezumab-Post-Treatment Phase: 300mg of galcanezumab given as SQ injections once every 28 days during a 12 week treatment period.
Arm/Group | Placebo - Treatment Phase | 5mg Galcanezumab-Treatment Phase | 50mg Galcanezumab-Treatment Phase | 120mg Galcanezumab-Treatment Phase | 300mg Galcanezumab-Treatment Phase | Placebo - Post-Treatment Phase | 5mg Galcanezumab-Post-Treatment Phase | 50mg Galcanezumab-Post-Treatment Phase | 120mg Galcanezumab-Post-Treatment Phase | 300mg Galcanezumab-Post-Treatment Phase
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/68 | 0/68 | 1/70 | 1/67 | 0/125 | 1/61 | 0/66 | 0/63 | 1/65
Other Adverse Events (participants affected / at risk) | 23/137 | 20/68 | 18/68 | 23/70 | 19/67 | 6/125 | 2/61 | 2/66 | 2/63 | 3/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=137) | 5mg Galcanezumab-Treatment Phase (N=68) | 50mg Galcanezumab-Treatment Phase (N=68) | 120mg Galcanezumab-Treatment Phase (N=70) | 300mg Galcanezumab-Treatment Phase (N=67) | Placebo - Post-Treatment Phase (N=125) | 5mg Galcanezumab-Post-Treatment Phase (N=61) | 50mg Galcanezumab-Post-Treatment Phase (N=66) | 120mg Galcanezumab-Post-Treatment Phase (N=63) | 300mg Galcanezumab-Post-Treatment Phase (N=65)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankyloglossia Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Following database lock, an additional SAE, ankyloglossia congenital, in a male infant of a paternal pregnancy case, was reported in the Lilly Safety System database (the father was treated with the 300-mg dose of galcanezumab).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Treatment Phase (N=137) | 5mg Galcanezumab-Treatment Phase (N=68) | 50mg Galcanezumab-Treatment Phase (N=68) | 120mg Galcanezumab-Treatment Phase (N=70) | 300mg Galcanezumab-Treatment Phase (N=67) | Placebo - Post-Treatment Phase (N=125) | 5mg Galcanezumab-Post-Treatment Phase (N=61) | 50mg Galcanezumab-Post-Treatment Phase (N=66) | 120mg Galcanezumab-Post-Treatment Phase (N=63) | 300mg Galcanezumab-Post-Treatment Phase (N=65)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (6) | 7 (11) | 6 (15) | 10 (13) | 9 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 8 (8) | 3 (3) | 6 (6) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 12 (15) | 7 (7) | 8 (8) | 8 (8) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (4) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days